CLINICAL TRIAL: NCT05720520
Title: Effect of Game-Based Virtual Reality Phone Application on Nursing Students' Knowledge and Skills on Intestinal Stoma and Peristomal Skin Care
Brief Title: Effect of Game-Based Phone Application on Nursing Students' Knowledge and Skills on Intestinal Stoma and Peristomal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Çalışkan, Research Assisstant, Abant Izzet Baysal University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: AIBU-SBF-MAC-02
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Nursing Education; Nursing Student; Phone Application; Stoma Care; Peristomal Skin Care; Virtual Reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Group (Experimental): Participants will use mobile application
  Interventions: Other: Technological education method
- Control Group (No Intervention): Participants only will take traditional education method

INTERVENTIONS:
Other: Technological education method — Students in the experimental group will play the mobile application developed for stoma and peristomal skin care and are expected to learn the skill in this way. The students in the control group, on the other hand, will learn stoma and peristomal skin care on a model in the traditional skill laboratory and are expected to learn the skill in this way. Afterwards, the knowledge and skill scores of the two groups will be compared and the results will be reported.
  Arms: Mobile Application Group

SUMMARY:
Purpose: The purpose is to determine effect of game-based virtual reality phone application on nursing students' knowledge and skills on intestinal stoma and peristomal skin care.

Material and methods:This study will be conducted as a single-blind randomized controlled experimental study between March-April 2023. The students in the experimental group will play the developed mobile game on stoma and peristomal skin care as much as they want for 5 days, while the students in the control group will perform skills on stoma and peristomal skin care on the model in the skill laboratory for only one day. After performing the inteventions, the skills and knowledge measurements of the students in both groups will be measured by the researcher through the forms prepared in accordance with the literature. After four weeks, the permanence levels of the students in both groups regarding stoma and peristomal skin care will be measured and the data collection process of the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* To register for the Nursing Fundamentals Course for the first time,
* Participating in theoretical lessons and group work,
* Participating in knowledge and skill assessments on stoma and peristomal skin care,
* Having an Android phone,
* Having internet access,
* Volunteer to participate in the research.

Exclusion Criteria:

* Have any previous training in stoma and peristomal skin care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Stoma and Peristomal Skin Care Skill Form | 1 day
  "Stoma and Peristomal Skin Care Skill Checklist" was prepared by the researcher in accordance with the literature. For the suitability of the skill checklist and scoring, the opinion of an expert in the field of Assessment and Evaluation, 10 faculty members who are experts in the field of Nursing Fundamentals in terms of content validity, and two specialist nurses working in the stoma and wound care unit were obtained by Davis Technique. The opinions of the experts were analyzed with the Lawshe technique and the Content Validity Index (CGI) of the form was found to be 0.98. Then, necessary arrangements were made in line with the recommendations of the experts.
  The checklist was classified as "Failed to perform" (0 points), "Partly performed" (1 point) and "Performed correctly" (2 points). "Stoma and Peristomal Skin Care Skill Checklist" consists of 27 steps and the lowest score that can be obtained from the scale is 0 and the highest score is 54. Higher scores indicate better results

SECONDARY OUTCOMES:
Stoma and Peristomal Skin Care Knowledge Form | 1 day
  The knowledge test was prepared by the researcher in accordance with the literature. The knowledge test is a test that questions students' knowledge of stoma and peristomal skin care. This test consists of 20 questions with five options. Each correct answer corresponds to 5 points. The lowest score 0 and the highest score 100 can be obtained from this test. Higher scores indicate better results. For the assurance of giving and obtaining information, an expert in the field of Assessment and Evaluation was obtained with the Davis technique, with 10 experts in the field of Nursing fundamentals in terms of the scope and validity of the scope. The opinions of the experts were analyzed with the Lawshe technique and the Scope Agreement Index (CGI) of the form was found to be 0.92. Necessary measures have been taken to ensure the training of trainers.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal Univercity, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No